CLINICAL TRIAL: NCT07392723
Title: Alpha Linolenic Acid-enriched Nutrition for Prevention of Cognitive Decline in APOE4 Older Adults With Mild Cognitive Impairment: Targeting Cerebrovascular and Blood-brain Barrier Health
Brief Title: ALA-enriched Nutrition for Prevention of Cognitive Decline in APOE4 Older Adults
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michal Schnaider Beeri, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Michal Schnaider Beeri, Ph.D., Krieger-Klein Endowed Chair in Neurodegeneration Research; Director of Herbert and Jacqueline Krieger Alzheimer's and Dementia Clinical Research and Treatment Center; and Professor of Neurology at Robert Wood Johnson Medical School, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro2025000006
Record Dates: First submitted 2025-10-20; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Dysfunction; Alzheimer Disease; Blood-Brain Barrier; Apolipoprotein E, Deficiency or Defect of; Brain Aging; Fatty Acids, Omega-3
Keywords: Alpha-Linolenic Acid; Flaxseed Oil; Apolipoprotein E4; Nutritional Intervention; APOE4 Dysfunction; Cognitive Function; Brain MRI; Blood Biomarkers; Vascular Integrity; Neurodegeneration; Aging Brain; Memory Loss Prevention; AD Prevention Trial; Alzheimer's Disease; Cognitive decline prevention; Blood-brain barrier; Dementia prevention; Older adults; Biomarkers; Magnetic resonance imaging (MRI)
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Apolipoprotein E, Deficiency or Defect of; Nerve Degeneration | interventions — alpha-Linolenic Acid; Linseed Oil; Corn Oil

STUDY DESIGN:
Intervention Model Description: Two groups:
  1. Flaxseed oil (ALA 2.6 g/day)
  2. Placebo (corn oil, iso-caloric control)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, study coordinators, and investigators conducting assessments will not know which oil each participant receives.
  Randomization and labeling are handled by the Rutgers Clinical Research Center Pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ALA Group (Experimental): Participants receive flaxseed oil in 5 mL oral syringes containing 2.6g of ALA, taken daily for six months.
  Interventions: Drug: Alpha-Linolenic Acid (2.6 g/day)
- Placebo Control Group (Placebo Comparator): Participants receive corn oil without ALA (iso-caloric placebo) in 5 mL oral syringes that are identical in appearance to those containing ALA, taken daily for six months.
  Interventions: Dietary Supplement: Placebo Control Group

INTERVENTIONS:
Drug: Alpha-Linolenic Acid (2.6 g/day) — Participants in this group will take flaxseed oil that contains 2.6 grams of alpha-linolenic acid (ALA) each day for six months. The oil will be provided in 5 mL prefilled oral syringes prepared by the Rutgers Clinical Research Pharmacy. Participants will take one syringe daily in the morning with food. They may mix the oil with cold foods such as yogurt or applesauce but should not heat it.
  The ALA supplement is intended to improve cognitive and brain health by enhancing the body's natural production of DHA that supports blood-brain barrier integrity and brain function.
  Other Names: Flaxseed Oil, ALA
  Arms: ALA Group
Dietary Supplement: Placebo Control Group — Participants in this group will take corn oil that does not contain ALA. The oil will be provided in the same 5 mL prefilled oral syringes as the active supplement and will look, taste, and smell similar to the ALA oil. Participants will take one syringe daily in the morning with food for six months.
  The placebo is used to compare effects against the ALA supplement and to maintain blinding for both participants and study staff.
  Other Names: Corn Oil, Placebo Control
  Arms: Placebo Control Group

SUMMARY:
This randomized, double-blind, placebo-controlled pilot trial will evaluate the effects of alpha-linolenic acid (ALA) supplementation on cognitive function, blood-brain barrier integrity, and brain vascular health in older adults with mild cognitive impairment and APOE4 genotype. By targeting the endogenous synthesis of docosahexaenoic acid (DHA) through ALA supplementation, the investigators aim to overcome the limitations of direct DHA supplementation, particularly in APOE4 carriers who exhibit low brain DHA levels and impaired blood-brain barrier function. This innovative approach offers a safe, cost-effective, and easily implementable therapeutic strategy for older adults at high risk for Alzheimer's dementia, especially APOE4 carriers, addressing a critical need given the limited cognitive benefits and significant adverse events of current amyloid-clearing drugs in this population.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled pilot study will evaluate the effects of alpha-linolenic acid (ALA)-enriched nutrition on cognitive function, blood-brain barrier (BBB) integrity, and brain vascular health in a high-risk population of older adults with MCI and APOE4 genotype. Docosahexaenoic acid (DHA), a critical fatty acid for brain health, is synthesized from ALA. Despite previous research showing limited cognitive benefits from DHA supplementation, APOE4 carriers have low brain DHA levels. This deficiency may stem from impaired transport across the BBB and compromised BBB integrity. The investigators hypothesize that ALA supplementation will enhance endogenous DHA synthesis, leading to improved cognitive outcomes through increased brain levels of DHA and its metabolites, including eicosapentaenoic acid (EPA) and docosapentaenoic acid (DPA), and improved BBB and brain vascular integrity. The study will include 60 older adults with MCI who carry at least one APOE4 allele. Participants will be randomized to either daily supplementation of 2.6 grams of ALA or a placebo (corn oil) for six months. The specific aims will compare ALA and placebo on: 1) Cognition: The investigators hypothesize improvement in global cognition at 6 months in the ALA-treated group. Secondary outcomes will be episodic memory and executive functions. 2) Cerebral vasculature: The primary neurobiological outcome will be BBB integrity, assessed via MRI. The investigators hypothesize that the ALA group will exhibit reduced BBB leakage compared to placebo. Secondary measures will include cerebral blood flow, brain vascular reactivity, and white matter hyperintensities. 3) Blood Biomarkers: The investigators will measure blood biomarkers indicative of BBB integrity (including mfsd2a, s100B, and GFAP). The investigators expect lower levels of these markers in the ALA group at six months, reflecting improved BBB function. Additionally, the investigators will analyze in plasma ALA and its downstream pathway (DHA, EPA). Finally, to distinguish the specific effects of ALA on cerebral vascular integrity from ADRD processes, the investigators will also explore its effects on plasma p-tau 217 and Neurofilament Light. This pilot study will lay the groundwork for a larger multi-site RCT testing the cognitive, BBB, and cerebrovascular benefits of ALA supplementation in APOE4 carriers at risk for Alzheimer's dementia. With current amyloid-clearing drugs showing limited success in preventing or reversing dementia symptoms-especially among APOE4 carriers-this research has potential for high public health impact by offering a promising new, low cost, safe therapeutic avenue for older adults at high dementia risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Have amnestic Mild Cognitive Impairment (MCI) - memory problems that do not interfere with daily life.
* Carry at least one APOE4 gene allele (determined by a blood test).
* Be fluent in English or Spanish.
* Have a study partner (family member or friend) who can provide information about daily function.
* Have the ability to give informed consent and comply with study visits and procedures.

Exclusion Criteria:

* A diagnosis of dementia or any other brain disease that significantly affects thinking or memory (e.g., Alzheimer's disease, Parkinson's disease, schizophrenia, epilepsy, traumatic brain injury).
* History of stroke or other major neurological condition.
* Short life expectancy due to end-stage disease or other serious medical condition.
* Active cancer treatment that could interfere with study participation.
* Allergy or sensitivity to flaxseed oil or corn oil.
* Current use of flaxseed, flax oil, or fish oil supplements more than once per week.
* MRI contraindications, such as pacemakers, metallic implants, or severe claustrophobia.
* Current or past history of prostate cancer, regardless of remission status, OR a prostate-specific antigen (PSA) level > 20 ng/mL at screening.
* Use of experimental Alzheimer's treatments (e.g., amyloid monoclonal antibodies) unless on a stable regimen as confirmed by the treating physician.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-12 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in global cognitive (score) function | Baseline and 6 months
  Change in global cognition score from baseline to 6 months measured by an average of the z-scores across a broad cognitive battery, will be compared between ALA and placebo groups.
Change in Blood-Brain Barrier Integrity - Permeability of the BBB | Baseline and 6 months
  Blood-brain barrier (BBB) permeability will be assessed using the water exchange rate constant (Kw), derived from a validated motion-corrected diffusion-weighted pseudocontinuous arterial spin labeling (MCDW-pCASL) MRI sequence. Values will be extracted from whole-brain and region-specific areas, including hippocampus, dorsolateral frontal cortex, and parietal cortex. Changes from baseline to 6 months will be compared between ALA and placebo groups.
Levels of blood biomarkers of BBB Integrity | baseline and 6 months
  Changes in protein levels in serum of: mfsd2a, s100B, and Glial Fibrillary Acidic Protein (GFAP) indicative of BBB function. Changes from baseline to 6 months will be compared between ALA and placebo groups.

SECONDARY OUTCOMES:
Episodic Memory | Baseline and 6 months
  Changes in episodic memory scores - the average z-score of the immediate and delayed word recall task, and the word recognition task will be assessed. Changes from baseline to 6 months will be compared between ALA and placebo groups.
Executive Function | Baseline and 6 months
  Changes in executive function scores - the average z-score of: Trail Making Test Parts A and B, Digit Span Forward and Backward, Animal Fluency, and Vegetable Fluency assessments. Changes from baseline to 6 months will be compared between ALA and placebo groups.
Cerebral Blood Flow | Baseline and 6 months
  Changes in cerebral blood flow will be assessed by MRI sequence measured by PSeudo Continuous Arterial Spin Labelling Sequence (pCASL). Values will be extracted from whole-brain and region-specific areas: hippocampus, as well as parietal, superior temporal, dorsolateral prefrontal, and precuneus cortex. Changes from baseline to 6 months will be compared between ALA and placebo groups.
Brain Vascular Reactivity | Baseline and 6 months
  Changes in brain vascular reactivity measured by a EPI BOLD scan tracing a CO2 concentration. Changes from baseline to 6 months will be compared between ALA and placebo groups.
White Matter Hyperintensity (WMH) | Baseline and 6 months
  Changes in WMH volume will be assessed using 3D T2-FLAIR MRI. Changes from baseline to 6 months will be compared between ALA and placebo groups.
Alzheimer's Disease and Related Dementia (ADRD) Blood Biomarkers - Phosphorylated tau 217 (p-tau217) and Neurofilament Light (NfL) | Baseline and 6 months
  Changes in plasma levels of Phosphorylated tau 217 (p-tau217) and Neurofilament Light (NfL) will be assessed. Changes from baseline to 6 months will be compared between ALA and placebo groups.
Blood fatty acids markers | Baseline and 6 months
  Changes in plasma levels of fatty acids including ALA, DHA, and EPA will be analyzed by TLC-GC-MS. Changes from baseline to 6 months will be compared between ALA and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Beeri, PHD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers - Institute for Health, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share non-identifiable (no PHI) data with other investigators upon participants' approval.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be made available after the main results of the study are published. This is anticipated to occur in June 2028.
Access Criteria: Qualified researchers will be able to access de-identified individual participant data and supporting documents (such as the study protocol and statistical analysis plan) upon reasonable request. Access will be provided after publication of the main results, following approval by the study sponsor and completion of a data use agreement.